CLINICAL TRIAL: NCT01580644
Title: Bioavailability Study of Two Formulations of the Isopropyl Malonate Prodrug of GLPG0187 in Healthy Male Subjects
Brief Title: Bioavailability Study of Prodrug of GLPG0187 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0187-CL-104
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Period 1: formulation 1 oral solution (Experimental)
  Interventions: Drug: GLPG0187 prodrug
- Period 2: formulation 2 capsule (Experimental)
  Interventions: Drug: GLPG0187 prodrug
- Period 3: Selected formulation + food (Experimental)
  Interventions: Drug: GLPG0187 prodrug
- Period 4: Selected formulation at higher dose (Experimental)
  Interventions: Drug: GLPG0187 prodrug

INTERVENTIONS:
Drug: GLPG0187 prodrug

SUMMARY:
The purpose of this study is to evaluate the amount of GLPG0187 present in the blood (pharmacokinetics) after a single oral dose of the prodrug of GLPG0187 given to healthy subjects.

Two formulations of the GLPG0187 prodrug will be compared, as well as the effect of food and dose proportionality of the best formulation.

Furthermore, during the course of the study, safety and tolerability will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The amount of GLPG0187 in plasma over time after a single oral dose of either of 2 formulations of GLPG0187 prodrug
  To characterize the amount of GLPG0187 in plasma over time - pharmacokinetics (PK) - after a single oral dose of either of 2 formulations of GLPG0187 prodrug in healthy subjects

SECONDARY OUTCOMES:
The amount of GLPG0187 in plasma over time after a single oral dose of the best formulation of GLPG0187 prodrug with food
  To characterize the amount of GLPG0187 in plasma over time - pharmacokinetics (PK) - after a single oral dose of the selected formulation of GLPG0187 prodrug with food in healthy subjects
The amount of GLPG0187 in plasma over time after a single oral dose of the best formulation of GLPG0187 prodrug at a higher dose (with or without food)
  To characterize the amount of GLPG0187 in plasma over time - pharmacokinetics (PK) - after a single oral dose of the selected formulation of GLPG0187 prodrug at a higher dose (with or without food) in healthy subjects to evaluate dose proportionality
Number of adverse events
  To evaluate the safety and tolerability of prodrug of GLPG0187 after a single oral dose in healthy subjects in terms of the number of adverse events reported
Changes in vital signs as measured by heart rate, blood pressure and body temperature
  To evaluate the safety and tolerability of prodrug of GLPG0187 after a single oral dose in healthy subjects in terms of changes in vital signs as measured by heart rate, blood pressure and body temperature reported
Changes on 12-lead ECG measures
  To evaluate the safety and tolerability of prodrug of GLPG0187 after a single oral dose in healthy subjects in terms of changes in 12-ECG measures reported
Changes in physical exam measures
  To evaluate the safety and tolerability of prodrug of GLPG0187 after a single oral dose in healthy subjects in terms of changes in physical examination reported
Changes in blood and urine safety lab parameters
  To evaluate the safety and tolerability of prodrug of GLPG0187 after a single oral dose in healthy subjects in terms of the changes in blood and urine safety lab parameters assessed

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV; Eva Vets, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Antwerp, Belgium